CLINICAL TRIAL: NCT06516432
Title: Serum Lactate in the Application of Parasternal Blockade in Trans and Post Anesthetic Stages in Cardiac Surgery
Brief Title: Parasternal Blockade and Serum Lactate in Cardiac Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, GONZALEZ-OJEDA ALEJANDRO, Principal Investigator, Instituto Mexicano del Seguro Social
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Parasternal Blockade 2024
Record Dates: First submitted 2024-07-10; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Elective Cardiac Surgery
Keywords: Parasternal block; Cardiac surgery; Serum lactate

STUDY DESIGN:
Intervention Model Description: Patients will be classified into a case group with parasternal block and a control group without parasternal block, with a ratio of cases to controls of 1:1.
  In the case-control groups, patients with elevated serum lactate levels above 2 mmol/L and those who remained below this limit will be identified.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case group (Experimental): with parasternal block
  Interventions: Procedure: Parasternal block; Procedure: Requirement of total dose regarding fentanyl
- Control group (No Intervention): without parasternal block

INTERVENTIONS:
Procedure: Parasternal block — In the case-control groups, patients with elevated serum lactate levels above 2 mmol/L and those who remained below this limit will be identified.
  Arms: Case group
Procedure: Requirement of total dose regarding fentanyl — In case-control groups, obtain measurement of total postoperative fentanyl requirement.
  Arms: Case group

SUMMARY:
Serum lactate level is a key indicator of tissue perfusion. Parasternal blockade is associated with reduced postoperative inflammatory response by inhibiting stress response, leading to better outcomes. Elevated lactate levels help identify patients at risk of postoperative morbidity and mortality. This analytical cross-sectional study evaluated the association between parasternal blockade and serum lactate levels in patients undergoing elective cardiac surgery in 2022 at Specialty Hospital CMNO. Patients with and without parasternal block were compared for changes in serum lactate levels during and after anesthesia within the first 24 hours.

DETAILED DESCRIPTION:
Background: Serum lactate level is a crucial indicator of tissue perfusion. Parasternal blockade has been related to a reduction of the postoperative inflammatory response, by inhibition of the stress response, leading to a better prognosis. Increased lactate level is a useful parameter in the identification of patients at risk of postoperative morbidity and mortality.

Objective: To evaluate the association between parasternal blockade and serum lactate level in patients undergoing cardiac surgery, both trans and postanesthesia.

Materials and Methods: Analytical cross-sectional study in adult patients undergoing elective cardiac surgery during the year 2022 in Specialty Hospital CMNO, patients with and without application of parasternal block were analyzed, and it was associated with changes in serum lactate level trans and post anesthesia in the first 24 hours. Approval registration: R-2023-1301-024.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients older than 18 years
* Either sex
* ASA II-III
* Patients who underwent cardiac surgery with median sternotomy and use of cardiopulmonary bypass.

Exclusion Criteria:

* Patients with pre-existing conditions that could independently affect serum lactate levels.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum lactate measurement | 24 hours postoperative
  Elevated serum lactate levels above 2 mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Gonzalez, 3, Principal Investigator — IMSS
Locations (1):
- Centro Médico Nacional de Occidente, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu H, Emelife PI, Prabhakar A, Moll V, Kendrick JB, Parr AT, Hyatali F, Pankaj T, Li J, Cornett EM, Urman RD, Fox CJ, Kaye AD. Regional anesthesia considerations for cardiac surgery. Best Pract Res Clin Anaesthesiol. 2019 Dec;33(4):387-406. doi: 10.1016/j.bpa.2019.07.008. Epub 2019 Jul 17. PMID 31791558
- [Background] Bloc S, Perot BP, Gibert H, Law Koune JD, Burg Y, Leclerc D, Vuitton AS, De La Jonquiere C, Luka M, Waldmann T, Vistarini N, Aubert S, Menager MM, Merzoug M, Naudin C, Squara P. Efficacy of parasternal block to decrease intraoperative opioid use in coronary artery bypass surgery via sternotomy: a randomized controlled trial. Reg Anesth Pain Med. 2021 Aug;46(8):671-678. doi: 10.1136/rapm-2020-102207. Epub 2021 May 14. PMID 33990437
- [Background] Chen Y, Li Q, Liao Y, Wang X, Zhan MY, Li YY, Liu GJ, Xiao L. Preemptive deep parasternal intercostal plane block for perioperative analgesia in coronary artery bypass grafting with sternotomy: a randomized, observer-blind, controlled study. Ann Med. 2023;55(2):2302983. doi: 10.1080/07853890.2024.2302983. Epub 2024 Feb 20. PMID 38375661
- [Background] Wong HMK, Chen PY, Tang GCC, Chiu SLC, Mok LYH, Au SSW, Wong RHL. Deep Parasternal Intercostal Plane Block for Intraoperative Pain Control in Cardiac Surgical Patients for Sternotomy: A Prospective Randomized Controlled Trial. J Cardiothorac Vasc Anesth. 2024 Mar;38(3):683-690. doi: 10.1053/j.jvca.2023.11.038. Epub 2023 Nov 30. PMID 38148266
- [Background] Li JQ, Li ZH, Dong P, Liu P, Xu YZ, Fan ZJ. Effects of parasternal intercostal block on surgical site wound infection and pain in patients undergoing cardiac surgery: A meta-analysis. Int Wound J. 2023 Oct 17;21(2):e14433. doi: 10.1111/iwj.14433. Online ahead of print. PMID 37846438
- [Background] Wang D, Wang S, Wu J, Le S, Xie F, Li X, Wang H, Huang X, Du X, Zhang A. Nomogram Models to Predict Postoperative Hyperlactatemia in Patients Undergoing Elective Cardiac Surgery. Front Med (Lausanne). 2021 Dec 2;8:763931. doi: 10.3389/fmed.2021.763931. eCollection 2021. PMID 34926506
- [Background] Yang HH, Chang JC, Jhan JY, Cheng YT, Huang YT, Chang BS, Chao SF. Prognostic value of peak lactate during cardiopulmonary bypass in adult cardiac surgeries: A retrospective cohort study. Tzu Chi Med J. 2020 Feb 27;32(4):386-391. doi: 10.4103/tcmj.tcmj_215_19. eCollection 2020 Oct-Dec. PMID 33163386
- [Background] Zhou Y, Yang C, Jin Z, Zhang B. Intraoperative use of cell saver devices decreases the rate of hyperlactatemia in patients undergoing cardiac surgery. Heliyon. 2023 May 4;9(5):e15999. doi: 10.1016/j.heliyon.2023.e15999. eCollection 2023 May. PMID 37215823
- [Background] Seghrouchni A, Atmani N, Moutakiallah Y, Belmekki A, El Bekkali Y, Houssa MA. Does severe hyperlactatemia during cardiopulmonary bypass predict a worse outcome? Ann Med Surg (Lond). 2021 Dec 21;73:103198. doi: 10.1016/j.amsu.2021.103198. eCollection 2022 Jan. PMID 35070281
- [Background] Demir AZ, Ozgok A, Balci E, Karaca OG, Simsek E, Gunaydin S. Preoperative ultrasound-guided bilateral thoracic erector spinae plane block within an enhanced recovery program is associated with decreased intraoperative lactate levels in cardiac surgery. Perfusion. 2024 Mar;39(2):324-333. doi: 10.1177/02676591221140754. Epub 2022 Nov 21. PMID 36408617
- [Background] Abadi A, Cohen R. Evaluation of an Enhanced Recovery After Surgery Protocol Including Parasternal Intercostal Nerve Block in Cardiac Surgery Requiring Sternotomy. Am Surg. 2021 Dec;87(10):1561-1564. doi: 10.1177/00031348211024638. Epub 2021 Jun 23. PMID 34162242
- [Background] Schiavoni L, Nenna A, Cardetta F, Pascarella G, Costa F, Chello M, Agro FE, Mattei A. Parasternal Intercostal Nerve Blocks in Patients Undergoing Cardiac Surgery: Evidence Update and Technical Considerations. J Cardiothorac Vasc Anesth. 2022 Nov;36(11):4173-4182. doi: 10.1053/j.jvca.2022.07.025. Epub 2022 Jul 24. PMID 35995636
- [Background] Padala SRAN, Badhe AS, Parida S, Jha AK. Comparison of preincisional and postincisional parasternal intercostal block on postoperative pain in cardiac surgery. J Card Surg. 2020 Jul;35(7):1525-1530. doi: 10.1111/jocs.14651. Epub 2020 Jun 24. PMID 32579779
- [Background] Miao Q, Wu DJ, Chen X, Xu M, Sun L, Guo Z, He B, Wu J. Target blood pressure management during cardiopulmonary bypass improves lactate levels after cardiac surgery: a randomized controlled trial. BMC Anesthesiol. 2021 Dec 8;21(1):309. doi: 10.1186/s12871-021-01537-w. PMID 34879822
- [Background] Caruso TJ, Lawrence K, Tsui BCH. Regional anesthesia for cardiac surgery. Curr Opin Anaesthesiol. 2019 Oct;32(5):674-682. doi: 10.1097/ACO.0000000000000769. PMID 31356362